CLINICAL TRIAL: NCT06777901
Title: Randomized Controlled Trial of the Auryon Atherectomy System Used in Combination With Standard Balloon Angioplasty Versus Standard Balloon Angioplasty Alone Treating Infrapopliteal Lesions in Subjects With Critical Limb Ischemia
Brief Title: Auryon Atherectomy System With Standard Balloon Angioplasty Versus Standard Balloon Angioplasty Alone
Acronym: AMBITION BTK
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Angiodynamics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-RFT-A-01
Record Dates: First submitted 2025-01-07; First posted 2025-01-16 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-05

CONDITIONS: Peripheral Arterial Diseases
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Angioplasty, Balloon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Auryon Atherectomy System and Balloon Angioplasty (Experimental): Subjects will be treated with the Auryon Atherectomy System followed by Percutaneous Balloon Angioplasty
  Interventions: Device: Auryon Atherectomy System
- Balloon Angioplasty Only (Active Comparator): Subjects assigned to this treatment group will be treated with percutaneous balloon angioplasty only.
  Interventions: Device: Balloon Angioplasty

INTERVENTIONS:
Device: Auryon Atherectomy System — Auryon Atherectomy System is composed of a laser and catheter
  Arms: Auryon Atherectomy System and Balloon Angioplasty
Device: Balloon Angioplasty — Balloon Angioplasty alone
  Arms: Balloon Angioplasty Only

SUMMARY:
The goal of this clinical trial is to learn if the Auryon Atherectomy System with balloon angioplasty safe and effective in treating lower limb blockages. The main question it aims to answer is: Is treatment with Auryon Atherectomy System more effective than angioplasty alone in preventing death, amputation, revascularization and improving patency? Researchers will compare the Auryon Atherectomy System with balloon angioplasty to balloon angioplasty alone.

DETAILED DESCRIPTION:
Up to 1500 subjects who do not meet the inclusion/exclusion criteria for the randomized study may satisfy the eligibility criteria for, and be enrolled in, the observational study.

ELIGIBILITY:
Inclusion Criteria:

* Age of subject is ≥ 18.
* Estimated life expectancy ≥1 year.
* Subject is able and willing to comply with all assessments in the study.
* Subject has been informed of the nature of the study, agrees to participate, and has signed the approved consent form.
* Rutherford Category classification of 4 or 5 of the target limb.
* Subject is a suitable candidate for angiography and endovascular intervention in the opinion of the investigator or per hospital guidelines.

Angiographic Inclusion Criteria

* Target lesion that is located in a native, de novo infra-popliteal artery (extending from P3 of the popliteal artery to the margin of the ankle mortise).
* Target lesions(s) must be viewed angiographically and have 50-100% stenosis.
* Only a single lesion is included in the study per subject.
* The vessel segment distal to the target lesion must be patent all the way to the ankle, with no significant lesion (≥ 50% stenosis).
* Lesion length ≥50mm and ≤300mm.
* Intraluminal crossing of the lesion. Successful crossing is defined as tip of the guidewire distal to the target lesion in the absence of flow limiting dissections or perforations. If this is not certain, IVUS or OCT may be used to verify this at the operator's discretion.
* Target Lesion reference vessel diameter (RVD) between 1.5mm - 4.5mm by investigator estimate.

Exclusion Criteria:

* Target lesion is in a vessel graft or synthetic graft.
* Treatment of target lesion with radial access.
* Planned target limb major amputation (above-the-ankle).
* Acute limb ischemia or required thrombolysis as a primary treatment modality of the target limb.
* History of prior endovascular or surgical procedure on the index limb within 30 days prior to enrollment or planned within 30 days of the index procedure.
* Subject is pregnant or breastfeeding. (Female subjects of childbearing potential must be non-breastfeeding and have a negative pregnancy test ≤ 7 days before the procedure.)
* Subject has a known coagulopathy or has bleeding diatheses/disorder, thrombocytopenia with platelet count less than 100,000/microliter / less than 80,000K.
* Subject in whom antiplatelet or anticoagulant therapy is contraindicated.
* Subject has known allergy to contrast agents or medications used to perform endovascular intervention that cannot be adequately pre-treated.
* Myocardial infarction within 60 days prior to enrollment.
* History of stroke/CVA/TIA within 60 days prior to enrollment.
* History of thrombolytic therapy within 14 days of enrollment.
* Subject has acute or chronic renal disease defined as serum creatinine of >2.5 mg/dL or >220 umol/L, or is on dialysis.
* Subject is participating in another research study involving an investigational agent (pharmaceutical, biologic, or medical device) that has not reached the primary endpoint.
* Subject has other medical, social or psychological problems that, in the opinion of the investigator, preclude them from receiving this treatment, and the study requirements and evaluations pre- and post-treatment.
* Subject experiencing ongoing cardiac problems that per the investigator judgment would not make the subject ideal per the procedure.
* Subject has evidence of intracranial or gastrointestinal bleeding within the past 3 months.

Angiographic Exclusion Criteria

* Failure to treat clinically significant inflow lesions in the ipsilateral iliac, femoral, or P1-P2 segments of the popliteal arteries with <50% residual stenosis with no serious angiographic complications (e.g., embolism or dissection) prior to treatment of the target lesion.
* Residual stenosis, and/or serious angiographic complications (e.g., embolism) prior to the investigational device usage.
* The use of adjunctive devices to treat the target lesion other than the investigative Auryon laser catheter and/or PTA devices, such as scoring balloons, drug-eluting balloons, re-entry devices, lithotripsy devices, or other atherectomy devices (with the exception of bailout stents for Class C/D dissections).

Subjects that do not meet eligibility criteria for the randomized controlled trial are eligible to be enrolled in the observational study.

Observational Study Inclusion Criteria:

* Subjects intended to be treated with the Auryon Atherectomy System for de-novo, restenotic or ISR lesions of the infra-popliteal arteries.
* Subjects presenting with symptomatic PAD with claudication or CLI by Rutherford Category 2 - 6 of the target limb.
* Age of subject is ≥ 18.
* Subject has been informed of the nature of the study, agrees to participate, and has signed the approved study consent form.

Observational Study Exclusion Criteria:

* Subjects with any medical condition that would make him/her an inappropriate candidate for treatment with Auryon Atherectomy System as per Instructions for Use (IFU) or investigator's opinion.
* Subject is pregnant or breastfeeding. (Female subjects of childbearing potential must be non-breastfeeding and have a negative pregnancy test ≤ 7 days before the procedure.)
* Subject is already enrolled in other investigational (interventional) studies that would interfere with study endpoints.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Win-ratio comparing subjects in the treatment group versus the control group on the components of the composite endpoints in a hierarchical fashion at 12 months | From enrollment to the end of treatment at 12 months
  The primary endpoint will be analyzed based on a Finkelstein-Schoenfeld/win-ratio approach, comparing pairs of subjects on the components of the composite endpoint in a hierarchical fashion:
  1. Freedom from amputation
  2. Freedom from CD-TLR
  3. Primary Patency

SECONDARY OUTCOMES:
Device Success | Measured upon completion of the index procedure
  Successful delivery, lesion crossing, functionality and retrieval of the investigational device
Procedural Success | Measured upon completion of the index procedure
  Defined as device success and residual diameter stenosis ≤30% on completion angiography without flow-limiting dissection (≥ grade D), perforation or distal embolization, all assessed by core lab on angiography.
Clinical Success | Measured upon completion of the index procedure prior to discharge.
  Defined as procedural success without procedural complications (death, major target limb amputation, thrombosis of the target lesion or TLR) prior to discharge.
Secondary Duplex Ultrasound Imaging Measures | Measured at Hospital Discharge (12-24 hours post-procedure or prior to discharge, whichever comes first), 30 days, and 6, 12, 24 months
  Subsegmental analysis: proportion of segments with binary restenosis (diameter stenosis of >50% or PSVR ≤ 2.5) on core lab-adjudicated DUS.
Primary sustained clinical improvement | Measured at 30 days, and 6, 12, 24 months
  Defined as freedom from target limb major amputation, CD-TLR and increase in Rutherford category from baseline.
Secondary Sustained Clinical Improvement | Measured at 30 days, and 6, 12, 24 months
  Defined as freedom from target limb major amputation and increase in Rutherford category from baseline.
Major Amputation | Measured at 30 days, and 6, 12, 24 months
  Defined as above-the-ankle amputation of the target limb.
Amputation-free survival | Measured at 30 days, and 6, 12, 24 months
  Defined as freedom from all-cause mortality and major amputation.
Primary Assisted Patency | Measured at 30 days, and 6, 12, 24 months
  Defined as freedom from Duplex ultrasound core laboratory (DCL)-adjudicated loss of patency (defined as ≥50% stenosis) irrespective of interventions for stenoses intended to maintain functionality and patency (defined as stenosis ≤50%)
Secondary Patency | Measured at 30 days, and 6, 12, 24 months
  Defined as freedom from loss of patency (defined as ≥50% stenosis) as determined by the DCL irrespective of interventions for stenoses intended to reestablish functionality and patency (defined as stenosis ≤50%
Clinically Driven Target Vessel Revascularization (CD-TVR) | Measured at 30 days, and 6, 12, 24 months
  Defined as re-intervention on target vessel due to recurrent/persistent/worsening symptoms and the Duplex ultrasound finding of ≥ 50% restenosis of target vessel by DCL measurement.
Rutherford Caregory | Measured at 30 days, and 6, 12, 24 months
  Defined as change in Rutherford category (0 asymptomatic -6 major tissue loss) from baseline.
Ankle Brachial Index/Toe-Brachial Index | Measured at 30 days, and 6, 12, 24 months
  Defined as change in Ankle-Brachial Index (ABI), or if unevaluable, Toe-Brachial index (TBI) from baseline.
Quality of Life (QOL) | Measured at 30 days, and 6, 12, 24 months
  Defined as change in Quality of Life (QOL) measures from baseline:
  - Walking Impairment Questionnaire (WIQ) - Defined as change in walking impairment questionnaire (WIQ) measures from baseline.
Rate of Major Adverse Limb Events | Measured at 30 days, and 6, 12, 24 months
  Defined as the composite of major amputation or major reintervention (new bypass graft, jump/interposition graft revision, thrombectomy/thrombolysis) of the index limb.
Rate of major cardiovascular event | Measured at 30 days, and 6, 12, 24 months
  Defined as the composite of cardiovascular death, myocardial infarction (MI), and stroke.
All-Cause Mortality | Measured at 30 days, and 6, 12, 24 months
Wound Healing | Measured at 30 days, and 6, 12, 24 months
  Defined as investigator-reported status of each index wound compared to baseline. Descriptive categories to be captured: 1) Improved 2) Unchanged 3) Worse 4) Healed/Complete Closure
Wound, Ischemia, foot Infection (WIfI) Classification | Measured at Discharge, 30 days, and 6, 12, 24 months
  Defined as the change in total WIfi score from baseline
Bailout Stenting | Measured upon completion of the index procedure prior to discharge.
  Bailout stenting will be allowed for: 1) flow-limiting Class C/D dissections or vessel perforations that are not amenable to two prolonged balloon inflations (≥ 2 min each); 2) acute vessel recoil or other negative occlusive complication that results in severely decreased vessel blood flow; or 3) persistent residual stenosis ≥30% by visual estimate after multiple prolonged balloon inflations.
Intravascular Imaging (IVI) analysis | Measured during the index procedure
  - Vessel calcification will be graded by IVI at baseline using the Fanelli classification.
Quality of Life (QOL) | Measured at 30 days, and 6, 12, 24 months
  Defined as change in Quality of Life (QOL) measures from baseline:
  - EQ-5D - Defined as change in health-related quality of life, encompassing five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Intravascular Imaging (IVI) analysis | Measured during the index procedure
  - Minimal luminal area (MLA) gain at the lesion site will be measured by IVI and calculated between after vessel prep prior to intervention, post-laser and post-PTA in the treatment arm, and after vessel prep prior to intervention and post-final adjunctive therapy in the control arm.
Intravascular Imaging (IVI) analysis | Measured during the index procedure
  - Dissections on IVI images will be classified using the iDissection classification

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Abrazo Arizona Heart Hospital, Phoenix, Arizona
  - Kaiser Permanente, San Diego, California
  - CIS Grey ASC, Gray, Louisiana
  - MedStar Health Research Institute, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Washington University, St Louis, Missouri
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Prisma Heath-University Medical Group, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: No